CLINICAL TRIAL: NCT04280107
Title: Evaluation of Styloid Chain Calcification to the Patient With the Temporomandibular Joint Disorder: a Retrospective Uncontrolled Cohort Study
Brief Title: Evaluation of Styloid Chain Calcification to the Patient With the Temporomandibular Joint Disorder
Status: Completed | Type: Observational
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Hatice Cansu Kış, Assistant Professor, Nuh Naci Yazgan University
Other Study IDs: 2018-615
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Styloid-Stylohoid Syndrome; Temporomandibular Disorder
Keywords: magnetic resonance imaging; cone beam computed tomography; temporomandibular dysfunction; Styloid-Stylohoid Syndrome
MeSH Terms: conditions — Eagle syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temporomandibular Dysfunction: For this study, 154 patient files who were admitted to the radiology department of the faculty of dentistry between 2013 and 2019 with complaints such as TMJ pain, mouth opening restriction, joint sound, joint function disorder were scanned retrospectively. Inclusion criteria: TMD patients with MR and CBCT images recorded in the digital archive. Exclusion criteria: Patients who have been operated or treated from TMJ, patients with head and neck trauma, patients with orthodontic treatment.

SUMMARY:
The aim of the study was to evaluate any relation between elongated styloid process (ESP) and type of Temporomandibular Joint Disorders (TMD).

DETAILED DESCRIPTION:
The styloid process (SP) of the temporal bone is a long conical cartilaginous projection lies anterior to the mastoid process. Patients who have ESP or styloid chain calcification are usually asymptomatic, only 4% are symptomatic. Symptoms vary as different syndromes which related affected anatomic structures by calcified process or ligament. Temporomandibular Dysfunction (TMD) describe the temporomandibular joint (TMJ) disfunction that divided three branches according to temporomandibular joint's disc status: non-displacement (ND), displacement with reduction (DWR) and displacement without reduction (DWoR). Since orofacial pain shows similar features in both ESP or styloid chain calcification and TMD, it is possible to confuse and misdiagnosis both of these clinical conditions. This study aimed to investigate the length and calcification pattern of the styloid process in patients with TMD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Temporomandibular Dysfunction(TMD)
* TMD patients with MR and CBCT images recorded in the digital archive.

Exclusion Criteria:

* operated or treated for any Temporomandibular Joint Diseases
* head and neck trauma
* orthodontic treatment

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have at least one of these clinic conditions: TMJ pain, mouth opening restriction, joint sound, joint function disorder.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Styloid chain calsifiaction pattern | 2 months
  Interpretation of Styloid chain calsifiaction pattern on reconstructed sagittal slices of CBCT.
Styloid processes length | 2 months
  Styloid processes length measured linearly on reconstructed sagittal slices of CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan, Turkey (Türkiye)

REFERENCES:
- [Derived] Kis HC, Soydan Cabuk D. Evaluation of styloid chain calcification related to temporomandibular joint disc displacement: a retrospective cohort study. Oral Radiol. 2021 Jul;37(3):395-402. doi: 10.1007/s11282-020-00463-w. Epub 2020 Jul 6. PMID 32632703